CLINICAL TRIAL: NCT04905901
Title: Does Nebulized Tranexamic Acid Affect Operative Field in Sinus Surgery? A Double Blind Randomized Clinical Trial
Brief Title: Nebulized Tranexamic Acid in Sinus Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Egypt Assuit university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300595
Record Dates: First submitted 2021-05-17; First posted 2021-05-28 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Bleeding Nose
MeSH Terms: conditions — Epistaxis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tranexamic acid 500 mg (Experimental): Nebulized tranexamic acid 500 mg 15 minutes before operation
  Interventions: Drug: Tranexamic acid
- Tranexamic acid 1gm (Experimental): Nebulized tranexamic acid 1 gm 15 minutes before operation
  Interventions: Drug: Tranexamic acid
- Saline placebo (Placebo Comparator): Normal saline nebulization 15 minutes before operation
  Interventions: Other: Saline placebo

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid nebulization 15 minutes before sinus surgery
  Other Names: Cyclokapron
  Arms: Tranexamic acid 1gm; Tranexamic acid 500 mg
Other: Saline placebo — Normal saline placebo nebulization 15 minutes before sinus surgery
  Arms: Saline placebo

SUMMARY:
The results of several recent studies on endoscopic sinus surgery through topical administration of tranexamic acid are encouraging in terms of the efficacy of tranexamic acid for intraoperative bleeding and other pathological conditions.The purpose of this study is to analyze the efficacy of nebulized tranexamic acid to improve the surgeon and patient experiences of sinus surgery and know the effective and safe dose of nebulized tranexamic acid.

DETAILED DESCRIPTION:
A written informed consent will be taken from the patients.The study involved adults of either sexes (age 18-65 years) of ASA I-II who will be listed for elective functional endoscopic sinus surgery (FESS) under general anesthesia, with normal accepted coagulation profile and hematocrit value ≥30 %. Excluded from the study patients with chronic renal failure, liver cirrhosis, bleeding disorders, current anticoagulant therapy, pregnancy or breastfeeding, impaired color vision, severe vascular ischemia, history of venous thrombosis, pulmonary embolism, long term treatment with acetylsalicylic acid or non-steroidal anti-inflammatory drugs not discontinued before surgery, a hemoglobin (HB) concentration <10 mg/dl or allergy to TXA.

Randomization: A random number sequence created by an internet website (http://www. random.org) will be used for patients' allocation. The random number sequence was retained in closed opaque envelopes released the day of the surgery by an independent physician not involved in the study. Patients will be assigned randomly to three groups (30 subjects each); saline placebo (Group S) and two different doses of preemptive nebulized tranexamic acid (Group T1) and (Group T2).To keep blinding, Group S will receive 2 sessions of nebulization each by 5 ml saline. Group T1 will receive one nebulization session 500 mg tranexamic acid (5 ml) and another one by 5 ml saline. Group T2 will receive 2 nebulization sessions each by 500 mg tranexamic acid (each by 5 ml)

ELIGIBILITY:
Inclusion Criteria:

* Either sexes (age 18-65 years) of ASA I-II who are listed for elective functional endoscopic sinus surgery (FESS) under general anesthesia
* normal accepted coagulation profile and hematocrit value ≥30

Exclusion Criteria:

* chronic renal failure
* liver cirrhosis
* bleeding disorders
* current anticoagulant therapy
* pregnancy or breastfeeding
* impaired color vision
* severe vascular ischemia
* history of venous thrombosis, pulmonary embolism
* long term treatment with acetylsalicylic acid or non-steroidal anti-inflammatory drugs not discontinued before surgery
* hemoglobin (HB) concentration <10 mg/dl _allergy to TXA.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
the Modena Bleeding Score (MBS) assessing surgical field | After anesthesia induction to 60 minute
  1= No bleeding, 2=Bleeding easily controlled by suctioning, washing or packing without any significant modification or slowing of surgical procedure, 3=Bleeding slowing surgical procedure, 4=Most of the maneuvers dedicated to bleeding control and 5=Bleeding that prevents every surgical procedure except those dedicated to bleeding control

SECONDARY OUTCOMES:
HR | Intraoperative duration
  Heart rate beat/min
MBP | Intraoperative duration
  Mean blood pressure mmHg
Anesthetic consumption | Anesthesia duration
  Extra doses of fentanyl and propofol and sevoflurane>2
Postoperative complications | After operation to 24 hour
  Recording any adverse effects to TXA e.g.nausea, vomiting and any visual disturbances

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided